CLINICAL TRIAL: NCT02018263
Title: Validation of a Remote Wireless Sensor Network (WSN) Approach to the Individualized Detection of Cocaine Use in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Gustavo Angarita, Assistant Professor of Clinical Psychiatry, Yale University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1212011268
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Cocaine; Exercise; Nicotine

ARMS (3):
- Cocaine Administration (Active Comparator): Subjects self administer cocaine hydrochloride in both laboratory and outpatient settings
  Interventions: Drug: Cocaine hydrochloride
- Nicotine Administation (Active Comparator): Subjects self administer nicotine in both laboratory and outpatient settings
  Interventions: Drug: Nicotine
- Exercise (Active Comparator): Subjects complete a cardiovascular exercise session in both laboratory and outpatient settings
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Drug: Cocaine hydrochloride
  Arms: Cocaine Administration
Behavioral: Exercise
  Arms: Exercise
Drug: Nicotine
  Arms: Nicotine Administation

SUMMARY:
This study looks to explore the feasibility, sensitivity, validity, and specificity of a Remote Wireless Sensor Network (RWSN) approach to the detection of cocaine use/intoxication in the inpatient human laboratory, as well as in the outpatient setting ("real world"). Lastly, we look to design an algorithm for reliably detecting cocaine use in real-world settings and inference techniques for understanding the relationship between cocaine use and user contexts.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 - 50 years,
2. voluntary, written, informed consent,
3. physically healthy by medical history, physical, neurological, ECG, and laboratory examinations,
4. DSM-IV criteria for Cocaine Abuse (305.60) or Cocaine Dependence (304.20)
5. recent street cocaine use in excess of amounts to be administered in the current study,
6. intravenous and/or smoked (crack/ freebase) use,
7. positive urine toxicology screen for cocaine,
8. for females, non-lactating, no longer of child-bearing potential (or agree to practice effective contraception during the study), and a negative serum pregnancy (β-HCG) test.

Exclusion Criteria:

1. Other drug dependence (except nicotine) as determined by urine toxicology or interview
2. < 1 year of cocaine dependence,
3. a primary major DSM-IV psychiatric diagnosis (schizophrenia, bipolar disorder, etc.), unrelated to cocaine,
4. a history of significant medical (cardiovascular) or neurological illness, ie prior myocardial infarction, current active symptoms of cardiovascular disease / angina, evidence of cocaine-related cardiovascular symptoms, prior arrhythmias or need for cardiov ascular resuscitation, neurovascular events such as transient ischemic attacks, stroke, and/or seizures Parameters re: elevations in vital signs are now explicitly specified under "Safety features built into our one-day self-administration paradigm).
5. current use of psychotropic and/or potentially psychoactive prescription medication,
6. seeking treatment for drug abuse/dependence (for experimental cocaine component),
7. physical or laboratory (β-HCG) evidence of pregnancy.
8. current use of any medication (prescription or over-the-counter) determined to cause potential drug interactions by the study physicians.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Instantaneous Heart Rate and Heart Rate Variability | 4 weeks

SECONDARY OUTCOMES:
Instantaneous Respiration Rate | 4 Weeks
Hand-based/Foot-based Skin Conductance | 4 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States